CLINICAL TRIAL: NCT00371436
Title: Progressive Intervention Program for Tinnitus Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C4488-R
Record Dates: First submitted 2006-08-31; First posted 2006-09-04 (Estimated); Results first posted 2015-04-08 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2015-03

CONDITIONS: Hearing Loss; Tinnitus
Keywords: Counseling; Education; Evaluation studies; Quality of health care; Rehabilitation of hearing impaired; Triage
MeSH Terms: conditions — Hearing Loss; Tinnitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Progressive Audiologic Tinnitus Management (PATM) (Active Comparator): The program follows a five-level "progressive intervention" model that addresses the various needs of tinnitus patients in a systematic and hierarchical manner-from initial contact with a VA provider through long-term treatment.
  Interventions: Procedure: Progressive Audiologic Tinnitus Management
- Usual Care (UC) (Other): Typical audiologic care that would be received in a VA Audiology Clinic.
  Interventions: Procedure: Usual Care

INTERVENTIONS:
Procedure: Progressive Audiologic Tinnitus Management — The five levels of progressive intervention are: (1) triage; (2) audiologic evaluation; (3) group education; (4) tinnitus evaluation; and (5) individual management.
  Other Names: PATM
  Arms: Progressive Audiologic Tinnitus Management (PATM)
Procedure: Usual Care — Typical audiologic care that would be received in a VA Audiology Clinic.
  Other Names: UC
  Arms: Usual Care (UC)

SUMMARY:
The purpose of this multi-site randomized clinical study is to test a model treatment program in a VA Audiology clinic, to evaluate its efficacy, ease of implementation, and acceptability to audiologists.

DETAILED DESCRIPTION:
The 2004 VA Annual Benefits Report reveals that tinnitus is the third most common individual service-connected disability in veterans. As of September 30, 2005, there were 339,573 veterans who had been awarded a service connection for their tinnitus, with annual compensation amounting to over $418,000,000 (Office of Policy and Planning, VA Central Office). In addition to being a major expense for VHA, tinnitus is a health care problem that is inadequately addressed at most VA medical centers. We have developed a research-based model of tinnitus clinical management that is designed for efficient implementation in VA Audiology clinics. The objective of this study is to establish the model program at a VA Audiology clinic, and to evaluate its efficacy with veteran patients and its acceptability to audiologists.

The study is based at the NCRAR, and a prototype tinnitus management program will be established in the Audiology Clinic at the James A. Haley (Tampa) VA Medical Center. The program follows a five-level "progressive intervention" model that addresses the various needs of tinnitus patients in a systematic and hierarchical manner-from initial contact with a VA provider through long-term treatment. It is hypothesized that progressive intervention will result in a significant reduction in self-perceived tinnitus handicap relative to usual care.

A comprehensive web-based tinnitus training course for audiologists has been developed, as well as a patient tinnitus-information book that uses principles of low health literacy. Six audiologists at the Tampa VA are participating in the study, of which three were randomly selected to complete the training course as preparation to conduct each of five levels of progressive intervention: (1) triage; (2) audiologic evaluation; (3) group education; (4) tinnitus evaluation; and (5) individualized management. The other three audiologists have not received the training, and these "usual care" audiologists provide intervention that more closely typifies what is done at some VA medical centers.

Patients will be randomized to one of the two groups. All patients will complete outcomes questionnaires (Tinnitus Handicap Inventory [THI] and Veterans Short Form-36 health survey [SF-36V]) at baseline, immediately post-treatment and 6 months post treatment. Outcomes of the THI will be compared between the two groups of patients to test the hypothesis. Data from the SF-36V will be used in secondary outcomes analyses. Each of the six audiologists will be interviewed informally to determine their satisfaction with the tinnitus services that they provide, and how they feel they are meeting the needs of their patients. The three web-based-trained audiologists will provide formative data to the Co-PI on an ongoing basis to monitor and adjust the program to achieve the best possible outcomes.

Development and evaluation of this prototype program will establish its practical utility for addressing the tinnitus needs of veterans in a comprehensive, yet efficient, fashion. If the study shows that the program is effective, then the program could establish the standard for tinnitus management at all VA medical centers-meeting the needs of all veterans who have access to VA services.

ELIGIBILITY:
Inclusion Criteria:

Veterans who:

* Are outpatients at VA clinics in the vicinity of the James A. Haley VA Medical Center in Tampa, FL
* Have clinically significant tinnitus
* Have no significant language barrier
* Are capable of and willing to fulfill all study requirements

Exclusion Criteria:

* Subjects must be free from any medical conditions that would interfere with study participation, e.g. medically or surgically treatable otologic disease; end-stage renal, pulmonary, or cardiovascular disease
* Patients undergoing chemotherapy or radiation treatment
* Patients with severe psychiatric disorders

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2008-09; Primary Completion 2009-09 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James A Henry, PhD, Principal Investigator — VA Medical Center, Portland
Locations (2):
- United States (2):
  - James A. Haley Veterans Hospital, Tampa, Tampa, Florida
  - VA Medical Center, Portland, Portland, Oregon

REFERENCES:
- [Result] Henry JA, Zaugg TL, Myers PJ, Kendall CJ, Michaelides EM. A triage guide for tinnitus. J Fam Pract. 2010 Jul;59(7):389-93. No abstract available. PMID 20625568
- [Result] Myers PJ, Griest S, Kaelin C, Legro MW, Schmidt CJ, Zaugg TL, Henry JA. Development of a progressive audiologic tinnitus management program for Veterans with tinnitus. J Rehabil Res Dev. 2014;51(4):609-22. doi: 10.1682/JRRD.2013.08.0189. PMID 25144174

RESULTS

PARTICIPANT FLOW:
Groups:
- Tinnitus Progressive Management: Tinnitus Progressive Management: The program follows a five-level "progressive intervention" model that addresses the various needs of tinnitus patients in a systematic and hierarchical manner-from initial contact with a VA provider through long-term treatment. The five levels of progressive intervention are: (1) triage; (2) audiologic evaluation; (3) group education; (4) tinnitus evaluation; and (5) individual management.
Period: Overall Study
Arm/Group | Tinnitus Progressive Management | Usual Care
Started | 92 | 89
Completed | 58 | 68
Not Completed | 34 | 21

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tinnitus Progressive Management | Usual Care | Total
Number analyzed (Participants) | 92 | 89 | 181
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.0 (11.2) | 59.0 (10.5) | 57.5 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 89 | 87 | 176
Region of Enrollment [Number; unit: participants]
  United States | 92 | 89 | 181

OUTCOME MEASURES:

1. Primary Outcome: THI (Tinnitus Handicap Inventory)
Description: The THI (Tinnitus Handicap Inventory) is a statistically validated tinnitus questionnaire that provides an index score, ranging from 0 to 100, with higher scores reflecting greater self-perceived tinnitus handicap.
Time Frame: Baseline, 6 months
Population: The THI was completed by 58 of the 92 PATM patients at both baseline and 6 months. The THI was completed by 68 of the 89 Usual Care patients at both baseline and 6 months.
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- Arm 1: Tinnitus Progressive Management
  Tinnitus Progressive Management: The program follows a five-level "progressive intervention" model that addresses the various needs of tinnitus patients in a systematic and hierarchical manner-from initial contact with a VA provider through long-term treatment. The five levels of progressive intervention are: (1) triage; (2) audiologic evaluation; (3) group education; (4) tinnitus evaluation; and (5) individual management.
- Arm 2: Usual Care
  Usual Care: Typical audiologic care that would be received in a VA Audiology Clinic.
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 58 | 68
scores on a scale
  Baseline | 37.0 (24.3) | 43.0 (25.4)
  6 months | 33.0 (26.4) | 40.0 (27.6)

ADVERSE EVENTS:
Description: Serious and other [non-serious] adverse events were not collected or assessed as part of the study.
Arm/Group | Tinnitus Progressive Management | Usual Care
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes